CLINICAL TRIAL: NCT03445325
Title: Project LiGHT (Living Green and Healthy for Teens): A Novel Weight Management Program That Emphasizes the Benefits of a Healthy Lifestyle
Brief Title: Pre/Post Evaluation of Living Green and Healthy for Teens (LiGHT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Childhood Obesity Foundation (Other); Ayogo Health Inc. (Other); Public Health Agency of Canada (PHAC) (Other Government); Merck Canada Inc. (Industry); Pacific Blue Cross (Unknown); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Louise Masse, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H16-03090-a
Record Dates: First submitted 2018-02-06; First posted 2018-02-26 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Pediatric
Keywords: obesity; physical activity; nutrition; adolescents; gamification; sedentary activity
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LiGHT v2.1 (Experimental): Participants will be assigned the intervention (use of the parent or teen app for 4.5 months) and asked to use throughout the intervention period (all participants are assigned to the intervention arm and results will be analyzed pre- and post-intervention).
  Interventions: Behavioral: LiGHT v2.1

INTERVENTIONS:
Behavioral: LiGHT v2.1 — The LiGHT mobile program strives to support youth and their families to adopt lifelong healthy behaviours in four areas - eating, physical activity, recreational screen time and sleep - to foster healthy growth and development, to prevent chronic diseases and manage unhealthy weights.
  The program includes content that involve the family, and focus on behavioural therapy as well as dietary and physical activity patterns. LiGHT is intended to be engaging and fun, provide virtual and tangible rewards, and interact with participants multiple times per day. In addition, it will feature a mobile social support network and interaction with a live coach with specialized training in motivational interviewing to support youth/families in changing their health behaviours through messaging and phone calls.

SUMMARY:
This study is the first of three sub-studies aimed at evaluating the outcomes of Living Green, Healthy for Teens (LiGHT v2.1), an app for 13 to 17 year -olds and their families that is intended to help them shift from an unhealthy lifestyle toward better health habits in three areas: physical activity, nutrition and sedentary behaviours. This first evaluation has the following aims to: 1) describe reach; 2) determine utilization/adherence to strategies implemented in the app and predictors of utilization/adherence; 3) assess change in knowledge and lifestyles behaviours associated with obesity as well as assess mediators of behaviour change. As this is a formative evaluation, it will prospectively follow 500 families for 4.5 months.

DETAILED DESCRIPTION:
Living Green, Healthy for Teens (LiGHT v2) is an engaging online, individualized, gamified lifestyle management program for youth focused on initiating long-term behaviour-change in youth and their families in order to help them shift from an unhealthy lifestyle toward better health habits in three areas: physical activity, nutrition and sedentary behaviour. The program aims both to treat and prevent childhood obesity, as well as to mitigate increased risk for metabolic and non-metabolic complications associated with obesity in the short and long-term.

Because parents have been shown to be of primary importance in treating childhood obesity, LiGHT v2 will educate and engage parents as well as youth. Parents will receive separate but complementary content, intended to guide them as they shop for and prepare food and make behavioural changes within their families. The content for parents will be delivered using the same social software that facilitates peer-to-peer conversations with teen users (forums), but the channels will be gated, so teens and parents each have their own space. LiGHT v2's social features will help parents strategize and empathize with other families facing similar challenges.

The program will be evaluated using three separate study groups. This protocol describes the first of the three.

A sample of 1400 families (one parent and one child) recruited by an online web panel will be screened for eligibility (i.e., children aged 13-17 and their parents). Of these, it is expected that approximately 500 will meet our eligibility criteria and express an interest in enrolling in the study, and of these, about 50% will actually enroll in the study. This evaluation will use a prospective design that integrates pre- and post-evaluations. All families will be given access to LiGHT v2.1 to use from their home computer and prospectively followed for 4.5 months.

Parents will complete questionnaires at baseline and after 4.5 months, which assess behaviours, sociodemographics, mediators of behaviour change, and satisfaction with the app. Teens will complete questionnaires at baseline, and after 1 and 4.5 months, which assess behaviours, satisfaction with the app, mediators of behaviour change, and knowledge for recommendations for healthy behaviours.

Parent/child usage will also be monitored using web-analytic tools in order to understand how users interact with LiGHT.

ELIGIBILITY:
Inclusion Criteria:

* Youth participants must be between the ages of 13 and 17
* Youth participants and at least one of their parents must be literate in English
* Youth participants and at least one of their parents must be able to read at the grade 5 level or above
* Parent participants must have primary custody of the child participant
* Families must have a computer or mobile device and internet access at home

Exclusion Criteria:

* Youth participants must not have any health condition that restricts the amount or type of activity the participant can do
* Youth participants must not have any health condition that severely restricts the types of food the participant can eat
* Youth participants must not have a diagnosis of type I diabetes
* Youth participants must not have any reason (including cognitive, psychological, or physical limitations) that preclude them from being able to spend 20-30 minutes using a computer program that is written at a 5th grade reading level

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Reach | Baseline
  Survey questions will assess socio-demographic characteristics of families and will be compared against those who were invited to participate in the study (from a web-based panel) and families who typically register for weight-management centres in Canada.
Adherence | Ongoing for 4.5 months
  Web-analytic tools will track utilization of LiGHT components and all interactions with the program. Adherence will be calculated as cumulative number of feature-specific interactions per week (e.g., number of interactions with articles, number of interactions with social wall, etc.).
Change in health behaviour knowledge | Baseline and 4.5 months
  Survey questions (using a LiGHT-specific tool) will assess teens' knowledge of Canadian recommendations for healthy eating, physical activity, and sedentary behaviours. Knowledge will be reported as an aggregate knowledge score from 0 to 13 (a score of 0 indicates low knowledge and a score of 13 indicates high knowledge), as well as sub-score for each of the knowledge area (healthy eating, physical activity, and sedentary behaviours).
Change in physical activity behavior (teens) | Baseline and 4.5 months
  Survey questions will assess teens' physical activity behaviours, and change in physical activity will be computed based on a composite physical activity score. Teen physical activity will be assessed using a modified version of the Physical Activity Questionnaire for Children (PAC-Q), and scored as average minutes per day of moderate-vigorous physical activity.
Change in physical activity behavior (parents) | Baseline and 4.5 months
  Survey questions will assess parents' physical activity behaviours, and change in physical activity will be computed based on a composite physical activity score. Parent physical activity will be assessed using a modified version of the International Physical Activity Questionnaire Short Form (IPAQ-SF), and scored as average minutes per day of moderate-vigorous physical activity.
Change in sedentary behaviour | Baseline and 4.5 months
  Survey questions will assess teens' and parents' recreational screen time use (using the Take Action survey), and will be reported as the number of self-reported hours of recreational screen time per day.
Change in dietary behaviour | Baseline and 4.5 months
  Survey questions will assess teens' and parents' dietary behaviours, and be reported as average number of fruits and vegetables and sugar-sweetened beverages per day.

SECONDARY OUTCOMES:
Change in mediators of behaviour change | Baseline, 1 month, and 4.5 months
  Survey questions will assess teens' self-efficacy and motivation in changing the health behaviours targeted by LiGHT

OTHER OUTCOMES:
Functionality | 4.5 months
  Monthly satisfaction surveys will assess whether users like the program (e.g. was LiGHT fun, easy to use and intuitive, did it offer content to which they could relate and features they like) and whether they have suggestions for improvement

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Masse, PhD, Principal Investigator — University of British Columbia School of Population and Public Health
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No